CLINICAL TRIAL: NCT03103815
Title: Trial of Amivita in Amyotrophic Lateral Sclerosis: a Single-center, Single-blind, Self-controlled Clinical Trial
Brief Title: Trial of Amivita in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wujin People's Hospital (Other)
Collaborators: Nanjing 1718 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WJ2017001
Record Dates: First submitted 2017-04-01; First posted 2017-04-06 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis, survival, adverse event
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a self-controlled trial. All participants will receive treatment.
Masking Description: The evaluating investigators will be blinded to treatment assignment. Patients in our center, include those participate in the trial and those receive standard therapy, will be evaluated by clinicians who do not know the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Experimental group will receive Amivita.
  Interventions: Drug: Amivita

INTERVENTIONS:
Drug: Amivita — In each course, Amivita solution (500ml) will be administrated i.v. once daily for 4 weeks. After an interval of 2 weeks, the participants will be treated again. A total of 7 courses will be given,

SUMMARY:
The primary objectives of this study are to determine the safety and efficacy of Amivita, a compound of amino acids and vitamines in patients with Amyotrophic lateral sclerosis (ALS)ALS. The secondary objectives are to measure quality of life before and during intervention. This is a self-controlled clinical trial. Twenty patients in our ALS center who are already receiving riluzole or other treatments but the condition is worsening will receive treatment for 1o months. The evaluating investigators will be blinded to treatment assignment. Primary outcome measures will be adverse events, the ALS Functional Rating Scale-Revised (ALSFRS-R), and survival. Subjects will also be assessed at enrollment and at study end for weight loss, forced vital capacity (FVC), quality of life and grip strength.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disorder affecting upper and lower motor neurons. Survival is typically 2 to 5 years from symptom onset; death is usually from respiratory paralysis. Standard therapy is with Riluzole 100 mg/day, a FDA approved treatment for ALS that has a small effect on survival. There is a strong need for more effective therapies in ALS.

In our previous studies, we have shown that Amivita, a compound of amino acids and vitamines, is effective for neuronal injury (unpublished data). We have since then use this regimen to treat ALS patients. Our retrospective analysis (unpublished data) of the treated patient indicates that this regimen can slow down the progression of ALS.

We proposed a self-controlled clinical trial to study the safety and efficacy of Amivita. Secondary outcome measures include weight and quality of life. Twenty subjects in our ALS center who are already receiving riluzole will receive treatment for 12 months. The evaluating investigators will be blinded to treatment assignment. Primary outcome measures will be adverse events, the ALS Functional Rating Scale-Revised (ALSFRS-R), and survival. Secondary outcome measures include body weight, forced vital capacity (FVC), quality of life and grip strength.

The total study length from first enrolled subject will be approximately 6 months.

Participants in this study will be subjects with familial or sporadic ALS diagnosed as probable, or definite, according to the World Federation of Neurology El Escorial criteria. Diagnostic and Inclusionary/Exclusionary criteria will be clearly outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria

* Patients must be men or women between the ages of 18 and 70 years
* Patient is clinical definite or probable ALS by the hospitals listed in the protocol
* Women who are of child bearing potential must have a negative pregnancy test
* Willing to comply with the study visits
* Will not take riluzole during the study period
* Be able to sign informed consent document

Exclusion Criteria

* Myotonic dystrophy
* Myasthenia gravis
* Post-poliomyelitis syndrome
* Multifocal motor neuropathy with or without conduction block
* Hirayama disease
* Kennedy disease
* Hereditary spastic paraplegia
* Syringomyelia
* Spinal cord and brain stem tumors
* Paraneoplastic syndromes
* Severe liver or kidney disease disease
* Infection, severe diarrhea or vomiting
* Serious heart or lung diseases or malignant tumor history
* HIV infection
* Pregnancy or breastfeeding
* Have no ability to communicate
* Have participated in other clinical trials within 4 weeks
* Any form of substance abuse, psychiatric disorder, or other condition that, in opinion of the investigator, may interfere with the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-10-20 (Estimated); Study Completion 2018-10-20 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) score | 10 months
  The ALSFRS is a validated clinical rating scale that has been shown to accurately track progression of patients disability in ALS. Inclusion of assessment of ALSFRS-R score is an essential element of the ALS trial.
  design of ALS clinical trials
Adverse event | 10 months
  Significant adverse events in gastrointestinal and respiratory symptoms will be written in the adverse event log. Safety laboratory studies will be drawn and site investigators will be notified by their clinical laboratories if there are any changes in the chemistry and liver functions tests.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 10 months
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration, measured in liters. FVC is an sensitive test for ALS patient' muscle ability.
EQ-5D | 10 months
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple measure of health for clinical appraisal.

OTHER OUTCOMES:
Grisp strength | 10 months
  A simple measure of muscle ability.
body weigh | 10 months
  Body weigh loss is common for ALS patients and is a simple measure for clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Maoxin Yue, M.D, Principal Investigator — Wujing People's Hospital
Locations (1):
- Wujing People's Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided